CLINICAL TRIAL: NCT06789874
Title: Comparing the Efficacy of Intralesional Saline Versus 35% Trichloracetic Acid (TCA) Peel in the Treatment of Atrophic Acne Scars
Brief Title: To Compare the Efficacy of Intralesional Saline Versus 35% Trichloracetic Acid (TCA) Peel in the Treatment of Atrophic Acne Scars
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Kainat usman, Post Graduate Resident in Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheikhzayedmedicalcollege SZMC
Record Dates: First submitted 2025-01-11; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Atrophic Acne Scar; Atrophic Acne Scarring
Keywords: Acne scars; TCA peel; Intralesional saline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralesional Saline for acne scars (Group A) (Active Comparator): Intralesional Saline 5 to 10ml injected in the sacrs fortnightly for 3 months
  Interventions: Procedure: Intralesional Saline
- Topical Trichloracetic acid for acne scars(Group B) (Active Comparator): 35% trichloroacetic acid peel was applied to scars monthly for 3 months
  Interventions: Procedure: 35% trichloracetic acid peel

INTERVENTIONS:
Procedure: Intralesional Saline — Intralesional Saline injected in scars
  Arms: Intralesional Saline for acne scars (Group A)
Procedure: 35% trichloracetic acid peel — 35%Trichloracetic acid peel was applied to scars monthly for 3 months
  Arms: Topical Trichloracetic acid for acne scars(Group B)

SUMMARY:
This study aimed to compare the efficacy of intradermal normal saline versus trichloroacetic acid (TCA) in treating atrophic acne scars. Atrophic acne scars are a common and disfiguring complication, with limited research on the use of normal saline.

DETAILED DESCRIPTION:
Acne vulgaris is a common skin problem affecting adolescents and adults. It is the eighth most common skin disease globally, having a prevalence ranging from 35%-85%, with notable variations across different regions and age groups.A randomized controlled trial was conducted at the Dermatology Department, Sheikh Zayed Hospital, Rahim Yar Khan, from 1st April 2023 to 31st October 2023. 126 patients were enrolled. Scar grading was based on Goodman and Baron's Qualitative Scar Classification. The Observer Scar Assessment Scale (OSAS) was used by dermatologists. Patients rated their acne scars using the Visual Disease Severity Scale. Photographs were taken for comparison. Efficacy was defined as ≥50% improvement in the OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-50 years
* Clinically diagnosed patients of atrophic acne scars on face
* duration of more than 6 months
* no history of any procedural intervention in past 3 months

Exclusion Criteria:

* history of keloid, active acne, local infection, skin allergies, hypertrophic scarring, photosensitivity, or history of any comorbidities
* history of use of oral isotretinoin, OCPs, steroids or immunosuppressants
* pregnant or lactating females

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Observer Scar Assessment Scale | clinical assessment will be done monthly for 6 months
  efficacy was labelled as improvement on observer scar assessment scale by >50% compared to baseline. Patient's satisfaction was recorded as 'not satisfied' (VAS score of 1-5), 'Satisfied' (VAS score of 6-7), and 'very satisfied' (Vas score of 8-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Zayed Medical College/Hospital, Rahimyarkhan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No